CLINICAL TRIAL: NCT03991416
Title: Understanding Your Baby: A Universal Parenting Support Program Aiming at Increasing Danish First Time Parents' Abilities for Understanding and Meeting Their Infants' Needs
Brief Title: Understanding Your Baby: A Parallel Group Study of a Universal Parenting Support Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Nordea-fonden (Unknown)
Responsible Party: Principal Investigator, Mette Væver, PhD, Associate Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCPH 2019-02
Record Dates: First submitted 2019-02-28; First posted 2019-06-19 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: First-time Mothers and Their Partners
Keywords: Universal; Prevention; Parental competence; Socioemotional; Public health nurses
MeSH Terms: interventions — Postnatal Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Understanding Your Baby (Experimental): Understanding Your Baby plus postnatal care as usual
  Interventions: Behavioral: Understanding Your Baby
- Care As Usual (Active Comparator): Postnatal care as usual
  Interventions: Behavioral: Postnatal care as usual

INTERVENTIONS:
Behavioral: Understanding Your Baby — Research-based knowledge on the understanding and meeting of the baby's socioemotional needs is delivered to the parents systematically by public health visitors based on a manual, cue cards, and video clips at four time points from 1 to 10 months postpartum.
  Other Names: Forstaa din baby
  Arms: Understanding Your Baby
Behavioral: Postnatal care as usual — In accordance with Danish national guidelines, health visitors visit families during the infants first year of life, where they weigh and measure the infant. Further, they offer individual guidance and support regarding for instance feeding, sleeping, how to stimulate the infant, and the developmental stages that the infant goes through.
  Arms: Care As Usual

SUMMARY:
In Understanding Your Baby first-time parents receive research-based knowledge on how to interpret their infants' socioemotional needs based on their behavior, and how to meet their infants' socioemotional needs in accordance with their developmental stage. This information is delivered to parents at routine home visits by public health nurses, who are trained in the research base behind the program, and using cue cards and short video clips, which concretely exemplify how infants signal their socioemotional needs and inspire to positive activities between parents and their infants.

The aim of Understanding Your Baby is to support infant socioemotional development by increasing parents' abilities at perceiving, understanding, and responding to their infant's socioemotional signals. Evaluation is based on a parallel group study, with half of the participants receiving care as usual and half of the participants receiving care as usual and Understanding Your Baby. The primary outcome is parental sense of competence and secondary outcomes are parental stress and child socioemotional development.

ELIGIBILITY:
Inclusion Criteria:

* First-time mother or father/partner
* Singleton pregnancy
* Mother living together with the baby
* Mother living in the Danish municipalities of Køge, Hvidovre, Høje-Taastrup, Frederiksberg, Lolland, Holbæk, Næstved, Middelfart, Nyborg or Aalborg.
* Understands Danish or English

Exclusion Criteria:

* Under the age of 18 when the child is born

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1737 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal Parenting Competence | T4 (infant age 11-11.5 months)
  Maternal Parenting Competence is assessed via self-report using the Parenting Sense of Competence Scale (PSOC; Gibaud-Wallston, 1977).

SECONDARY OUTCOMES:
Maternal and Paternal Parenting Competence | T1 (infant age 2-2.5 months), T2 (infant age 4-4.5 months), and T3 (infant age 7-7.5 months)
  Maternal and paternal parenting competence is assessed via self-report using the Parenting Sense of Competence Scale (PSOC; Gibaud-Wallston, 1977).
Maternal and Paternal Parenting Stress | T2 (infant age 4-4.5 months) and T4 (infant age 11-11.5 months)
  Maternal and paternal parenting stress is assessed via self-report using the Parenting Stress Index™, Third Edition Short Form (PSI-3-SF; Abidin, 1995).
Maternal and Paternal Parental Mentalizing | T2 (infant age 4-4.5 months), T3 (infant age 7-7.5 months), and T4 (infant age 11-11.5 months)
  Maternal and paternal parental mentalizing is assessed via self-report using the Parental Reflective Functioning Questionnaire (PRFQ; Luyten, Mayes, Nijssens, & Fonagy, 2017).
Maternal and Paternal Mind-Mindedness | T1 (infant age 2-2.5 months), T2 (infant age 4-4.5 months), T3 (infant age 7-7.5 months), and T4 (infant age 11-11.5 months)
  Maternal and paternal mind-mindedness are assessed using a written response to the first question from the "Describe you child" interview (Meins et al., 1998). Mind-mindedness is coded according to the criteria specified in the mind-mindedness coding manual (Meins & Fernyhough, 2015).
Maternal, paternal and child screen use | T1 (infant age 2-2.5 months), T2 (infant age 4-4.5 months), T3 (infant age 7-7.5 months), and T4 (infant age 11-11.5 months)
  Maternal, paternal and child screen use is measured using a questionnaire developed specifically for this research project.
Infant socio-emotional development | T4 (infant age 11-11.5 months)
  Infant socio-emotional development is assessed via parental report using the Ages & Stages Questionnaires®: Social-Emotional, Second Edition (ASQ:SE-2; Squires, Bricker, & Twombly, 2015).

CONTACTS AND LOCATIONS:
Overall Officials: Mette S. Væver, Principal Investigator — University of Copenhagen
Locations (1):
- Center for Early Interventions and Family Studies, Department of Psychology, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaever MS, Krogh MT, Stuart AC, Madsen EB, Haase TW, Egmose I. Understanding Your Baby: protocol for a controlled parallel group study of a universal home-based educational program for first time parents. BMC Psychol. 2022 Sep 22;10(1):223. doi: 10.1186/s40359-022-00924-3. PMID 36138482